CLINICAL TRIAL: NCT02981134
Title: The Usefulness of Coronary CT Scan After Everolimus-eluting Bioabsorbable Scaffold Implantation for Coronary Artery Disease; A Single Center, Prospective Observational Study
Brief Title: The Usefulness of Coronary CT Scan After Everolimus-eluting Bioabsorbable Scaffold Implantation for Coronary Artery Disease
Acronym: CT BVS
Status: Withdrawn | Type: Observational
Why Stopped: This study will be revived with retrospective design.
Sponsor: Jung-min Ahn (Other)
Collaborators: CardioVascular Research Foundation, Korea (Other)
Responsible Party: Sponsor-Investigator, Jung-min Ahn, Assistant professor, Department of Cardiology, Heart Institute, University of Ulsan College of Medicine, Asan Medical Center
Organization: Asan Medical Center (Other)
Other Study IDs: AMCCV2016-25
Record Dates: First submitted 2016-11-30; First posted 2016-12-05 (Estimated); Last update posted 2021-07-23 (Actual); Status verified 2021-07

CONDITIONS: Coronary Disease
Keywords: bioabsorbable scaffold; computed tomography
MeSH Terms: conditions — Coronary Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- bioabsorbable scaffold: Patients with BVS(bioabsorbable scaffold) for coronary stenosis
  Interventions: Procedure: Computed tomographic scan

INTERVENTIONS:
Procedure: Computed tomographic scan — after 1year of BVS implantation, computed tomographic scan will be performed

SUMMARY:
The purpose of this study is to evaluate usefulness of coronary computed tomographic scan for prediction of clinical events after everolimus-eluting bioabsorbable scaffold implantation for coronary artery disease.

ELIGIBILITY:
Inclusion Criteria:

* Patients treated withBioresobable Vascular Scaffold for coronary disease

Exclusion Criteria:

* History of allergy to contrast
* Serum Creatinine > 2.0 mg/dl
* Severe arrhythmia
* Pregnancy or breast feeding

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients treated with Bioresobable Vascular Scaffold for coronary disease
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2021-12 (Estimated); Primary Completion 2023-06 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Computed tomographic scan parameters | 3 years
  Computed tomographic scan parameters predicting clinical outcomes

SECONDARY OUTCOMES:
Restenosis | 1 year
  Restenosis on computed tomographic scan
Thrombosis | 1 year
  Thrombosis on computed tomographic scan
Lumen loss | 1 year
  lumen loss: the change in minimal lumen diameter on computed tomographic scan
Positive predictive value | 3 years
  Positive predictive value on computed tomographic scan
Clinical outcomes | 3 years
  Death, target vessel myocardial infarction, clinically driven revascularization
Proportion of analyzable lesion | 3 years
  small vessel defined diameter less than 3.0 mm, bifurcation, overlapped lesion

CONTACTS AND LOCATIONS:
Locations (1):
- Asan Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided